CLINICAL TRIAL: NCT02474407
Title: An Open-Label, Randomized, Crossover Pharmacokinetic Study to Determine the Bioavailability, Safety and Tolerability of Single Doses of Diazepam Nasal Spray Versus Diazepam Rectal Gel (Diastat®) in Patients With Refractory Epilepsy
Brief Title: Bioavailability, Safety and Tolerability of Diazepam Nasal Spray Versus Diazepam Rectal Gel (Diastat®)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DZNS-EP-1019
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Refractory Epilepsy
Keywords: Seizures; Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures; Epilepsy | interventions — Diazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diazepam nasal spray (DZNS) (Experimental): One dose of diazepam nasal spray is administered as two intranasal sprays; one in each nostril using a nasal spray device.
  Interventions: Drug: diazepam nasal spray
- diazepam rectal gel (DRG) (Active Comparator): A single rectal dose of diazepam will be administered to subjects according to the Diastat prescribing information.
  Interventions: Drug: diazepam rectal gel

INTERVENTIONS:
Drug: diazepam nasal spray
  Other Names: Diazepam
  Arms: diazepam nasal spray (DZNS)
Drug: diazepam rectal gel
  Other Names: Diastat®; AcuDial™
  Arms: diazepam rectal gel (DRG)

SUMMARY:
This is a multi-center, open-label, crossover, pharmacokinetic, bio-availability study involving adolescents and adults with refractory (drug-resistant) epilepsy. Cohort 1 comprises the subjects used to determine the relative bioavailability of DZNS versus DRG (Diastat)

DETAILED DESCRIPTION:
To determine the bioavailability of diazepam nasal spray versus diazepam rectal gel (Diastat®) under conditions of use in adolescent and adult persons with epilepsy (PWE) meeting the definition of refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory epilepsy
* Body weight 26 to 111 kilogram (kg) inclusive
* Other inclusion criteria apply

Exclusion Criteria:

* Male or female subject who is not surgically sterile or female subject who is less than 2 years postmenopausal, and does not agree to use a highly effective birth control method during the study and up to 3 months after the last dose of investigational product
* Female subject who is pregnant, breastfeeding, or planning to become pregnant
* Presence or history of any abnormality or illness that may affect the absorption, distribution, metabolism or elimination of diazepam
* Other exclusion criteria apply

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Min Jae, Study Director — SK Biopharmaceuticals Co, Ltd
Locations (22):
- United States (22):
  - Acorda Site #115, Little Rock, Arkansas
  - Acorda Site #127, Washington D.C., District of Columbia
  - Acorda Site #101, Tampa, Florida
  - Acorda Site #125, Honolulu, Hawaii
  - Acorda Site #104, Lexington, Kentucky
  - Acorda Site #111, Baltimore, Maryland
  - Acorda Site #102, Bethesda, Maryland
  - Acorda Site #110, Ann Arbor, Michigan
  - Acorda Site #117, Jackson, Mississippi
  - Acorda Site #112, St Louis, Missouri
  - Acorda Site #128, Edison, New Jersey
  - Acorda Site #121, Hackensack, New Jersey
  - Acorda Site #123, Amherst, New York
  - Acorda Site #119, Rochester, New York
  - Acorda Site #132, Chapel Hill, North Carolina
  - Acorda Site #114, Portland, Oregon
  - Acorda Site #116, Philadelphia, Pennsylvania
  - Acorda Site #105, Philadelphia, Pennsylvania
  - Acorda Site #130, Memphis, Tennessee
  - Acorda Site #103, Bellaire, Texas
  - Acorda Site #122, Dallas, Texas
  - Acorda Site #108, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized crossover study with 78 subjects total.
Groups:
- Single Dose of Diazapam Nasal Spray (DZNS): Subjects received a single dose diazepam nasal spray (DZNS) followed by a washout period of 14 days, after which a single dose of diazapam rectal gel (DRG) was administered.
- Single Dose of Diazapam Rectal Gel (DRG): Subjects received a single dose of Diazepam Rectal Gel (DRG) followed by a washout period of 14 days, after which a single dose of diazapam nasal spray (DZNS) was administered.
Period: First Intervention (14 Days)
Arm/Group | Single Dose of Diazapam Nasal Spray (DZNS) | Single Dose of Diazapam Rectal Gel (DRG)
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Single Dose of Diazapam Nasal Spray (DZNS) | Single Dose of Diazapam Rectal Gel (DRG)
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Single Dose of Diazapam Nasal Spray (DZNS) | Single Dose of Diazapam Rectal Gel (DRG)
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: DZNS (Diazepam Nasal Spray) vs DRG (Diazepam rectal gel)
Arm/Group | All Participants
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 75
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 57
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-24h
Description: Relative bioavailability based on area under time plasma concentration curve.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Single Dose of Diazapam Nasal Spray (DZNS); Single Dose of Diazapam Rectal Gel (DRG): Single, weight-based dose (0.2mg/kg) of DZNS and DRG administered in two randomly assigned treatment periods, separated by a minimum 14-day washout period per intervention.
Arm/Group | Single Dose of Diazapam Nasal Spray (DZNS) | Single Dose of Diazapam Rectal Gel (DRG)
Number analyzed (Participants) | 78 | 78
ng*h/mL | 1357.7 (802.78) | 2117.9 (996.27)

2. Primary Outcome: Cmax
Description: Relative bioavailability based on maximum observed plasma concentration.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Single Dose of Diazapam Nasal Spray (DZNS) | Single Dose of Diazapam Rectal Gel (DRG)
Number analyzed (Participants) | 78 | 78
ng/mL | 157.0 (120.15) | 309.3 (137.95)

3. Secondary Outcome: Focused Nasal Exam (Part A)
Description: A focused nasal exam was completed by the Investigator in the treatment period(s) when diazepam nasal spray was administered, based on a visual inspection of the nasal mucosa. Nasal irritation will be graded "none" to Grade 4 "septal perforation." Grade 1a= focal irritation, Grade 1b= superficial mucosal erosion, Grade 2= moderate mucosal erosion, Grade 3= ulceration, Grade 4= septal perforation. This exam may be conducted within a 5 minute window after the specified time point. Between the 12 and 24 h time points, the exam should be repeated every 4 hours as needed to follow any residual symptoms to resolution and the time of resolution should be documented.
  (Categories with no data were omitted)
Time Frame: pre-dose (day 1) up to 24 hours post-dose
Population: Safety population Cohort 1. (Accessed only for DZNS Arm)
Measure: Count of Participants; unit: Participants
Groups:
- DZNS - At 24 Hours Post-Dose - NONE; DZNS - At 24 Hours Post-Dose - Grade 1a; DZNS - At 24 Hours Post-Dose - Grade 1b; DZNS - At 24 Hours Post-Dose - Grade 2; DZNS - At 24 Hours Post-Dose - Grade 3; DZNS - At 24 Hours Post-Dose - Grade 4; DZNS - At 24 Hours Post-Dose - Missing: One dose of diazepam nasal spray is administered as two intranasal sprays; one in each nostril using a nasal spray device.
  diazepam nasal spray
Arm/Group | DZNS - At 24 Hours Post-Dose - NONE | DZNS - At 24 Hours Post-Dose - Grade 1a | DZNS - At 24 Hours Post-Dose - Grade 1b | DZNS - At 24 Hours Post-Dose - Grade 2 | DZNS - At 24 Hours Post-Dose - Grade 3 | DZNS - At 24 Hours Post-Dose - Grade 4 | DZNS - At 24 Hours Post-Dose - Missing
Number analyzed (Participants) | 78 | 78 | 78 | 78 | 78 | 78 | 78
Participants
  Nasal Irritation at Baseline - NONE | 64 | 6 | 0 | 1 | 0 | 0 | 0
  Grade 1a | 1 | 3 | 0 | 0 | 0 | 0 | 0
  Grade 1b | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Focused Nasal Exam (Part B)
Description: A focused nasal exam was completed by the Investigator in the treatment period(s) when diazepam nasal spray was administered, based on a visual inspection of the nasal mucosa. Focused Nasal Examination Part B - will show nasal mucosal symptoms that will be rated for severity will include discharge, mucosal edema, crusting, erythema, and epistaxis. This exam may be conducted within a 5 minute window after the specified time point. Between the 12 and 24 h time points, the exam was should be repeated every 4 hours as needed to follow any residual symptoms to resolution and the time of resolution should be documented.
  (Categories with no data were omitted)
Time Frame: pre-dose (day 1) up to 24 hours post-dose
Population: The Safety population / Cohort 1. (Accessed only for DZNS Arm)
Measure: Count of Participants; unit: Participants
Groups:
- DZNS - At 24 Hours Post-Dose None; DZNS - At 24 Hours Post-Dose Mild; DZNS - At 24 Hours Post-Dose Moderate; DZNS - At 24 Hours Post-Dose Severe; DZNS - At 24 Hours Post-Dose Missing: One dose of diazepam nasal spray is administered as two intranasal sprays; one in each nostril using a nasal spray device.
  diazepam nasal spray
Arm/Group | DZNS - At 24 Hours Post-Dose None | DZNS - At 24 Hours Post-Dose Mild | DZNS - At 24 Hours Post-Dose Moderate | DZNS - At 24 Hours Post-Dose Severe | DZNS - At 24 Hours Post-Dose Missing
Number analyzed (Participants) | 78 | 78 | 78 | 78 | 78
Participants
  At Baseline: Mucosal Edema-None | 70 | 3 | 0 | 0 | 0
  Mucosal Edema - Mild | 1 | 3 | 0 | 0 | 0
  Mucosal Edema - Moderate | 0 | 1 | 0 | 0 | 0
  At Baseline: Nasal Discharge - None | 67 | 7 | 1 | 0 | 0
  Nasal Discharge - Mild | 1 | 1 | 0 | 0 | 0
  Nasal Discharge - Moderate | 0 | 1 | 0 | 0 | 0
  At Baseline: Mucosal Erythema - None | 67 | 6 | 0 | 0 | 0
  Mucosal Edrythema - Mild | 0 | 5 | 0 | 0 | 0
  At Baseline: Mucosal Bleeding/Epistaxis - None | 76 | 1 | 0 | 0 | 0
  Mucosal Bleeding/Epistaxis - Mild | 1 | 0 | 0 | 0 | 0
  At Baseline: Crusting of Mucosa - None | 77 | 1 | 0 | 0 | 0

5. Secondary Outcome: Smell Identification Test (SIT)
Description: The SIT is a validated test of smell identification which scores patients into different levels of olfactory function normalized by age and gender, however it had not been validated for use in PWE. The Smell Identification Test (SIT) is a 40-item multiple-choice standardized test. The test can be self-administered and consists of four 10-page booklets with a different "scratch and sniff" strip on each page. A scratch with a pencil releases the scent from the strip, and the subject is then asked to match the scent to one of four choices on the page. An answer must be selected for each of the 40 items, even when the subject cannot detect a smell. The total score (i.e., number of correct answers, range: 0-40) can be compared against normative data collected from approximately 4000 normal individuals between ages 4 to 99 to determine the subject's percentile rank of olfactory dysfunction corrected for age and gender.
Time Frame: day 1 up to day 31
Population: Safety Population / Cohort 1. (Accessed only for DZNS Arm)
Measure: Count of Participants; unit: Participants
Groups:
- At Follow-Up Visit - Normosmia; At Follow-Up Visit - Mild Microsmia; At Follow-Up Visit - Moderate Microsmia; At Follow-Up Visit - Severe Microsmia; At Follow-Up Visit - Anosmia; At Follow-Up Visit - Probable Malingering; At Follow-Up Visit - Missing: Shift in SIT Scores in Cohort 1 from Treatment Period 1 (Prior to Dosing) to Follow-up Visit
Arm/Group | At Follow-Up Visit - Normosmia | At Follow-Up Visit - Mild Microsmia | At Follow-Up Visit - Moderate Microsmia | At Follow-Up Visit - Severe Microsmia | At Follow-Up Visit - Anosmia | At Follow-Up Visit - Probable Malingering | At Follow-Up Visit - Missing
Number analyzed (Participants) | 78 | 78 | 78 | 78 | 78 | 78 | 78
Participants
  At BASELINE: Normosmia | 19 | 10 | 0 | 0 | 0 | 0 | 1
  Mild Microsmia | 2 | 10 | 5 | 1 | 0 | 0 | 0
  Moderate Microsmia | 2 | 3 | 3 | 6 | 1 | 0 | 0
  Severe Microsmia | 0 | 1 | 1 | 4 | 1 | 0 | 0
  Anosmia | 0 | 0 | 0 | 2 | 3 | 0 | 1
  Probable Malingering | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 2

6. Secondary Outcome: Taste Change Questionnaire
Description: Questionnaire given to safety population in Cohort 1 for reporting taste change during the study. If the subject spontaneously reports an experience of taste change associated with diazepam nasal spray dosing, it will be evaluated qualitatively by the research staff using a taste change questionnaire. The subject will be asked to describe the type, intensity, and duration of the change in taste at multiple scheduled time points after dosing. Between the 12 and 24 h time points, the questionnaire should be repeated every 4 hours as needed to follow any residual symptoms to resolution, and time of resolution should be documented.
Time Frame: Up to 24 hours
Population: Safety Population / Cohort 1. (Accessed only for DZNS Arm)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Taste Change by Intensity in Cohort 1: Questionnaire for taste change associated with diazepam nasal spray dosing.
Arm/Group | Taste Change by Intensity in Cohort 1
Number analyzed (Participants) | 78
units on a scale
  5 mins Post-Dose | 6.5 (3.57)
  15 mins Post-Dose | 4.6 (3.09)
  30 mins Post Dose | 2.8 (2.75)
  1 hr Post Dose | 1.0 (1.45)
  2 hrs Post-Dose | 0.3 (0.48)
  4 hrs Post-Dose | 0.1 (0.36)
  8 hrs Post-Dose | 0.0 (0.0)
  12 hrs Post-Dose | 0.0 (0.0)
  24 hrs Post-Dose | 0.0 (0.0)

ADVERSE EVENTS:
Time Frame: 31 Days
Groups:
- Diazepam Nasal Spray: One dose of diazepam nasal spray is administered as two intranasal sprays; one in each nostril using a nasal spray device.
  Diazepam Nasal Spray
- Diazepam Rectal Gel: A single rectal dose of diazepam will be administered to subjects according to the Diastat prescribing information.
  Diazepam Rectal Gel
Arm/Group | Diazepam Nasal Spray | Diazepam Rectal Gel
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 60/78 | 20/78
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diazepam Nasal Spray (N=78) | Diazepam Rectal Gel (N=78)
Nasal Discomfort (General disorders) | 30 | 3
Dysgeusia (General disorders) | 25 | 0
Lacrimation Increased (General disorders) | 22 | 0
Nasal Mucosal Disorder (General disorders) | 10 | 2
Rhinorrhea (General disorders) | 10 | 1
Edema Mucosal (General disorders) | 8 | 1
Throat irritation (General disorders) | 9 | 0
Somnolence (Nervous system disorders) | 4 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Headache (Nervous system disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Feeling Hot (General disorders) | 1 | 0
Mucosal erosion (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Secretion discharge (General disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
White blood cell count (Investigations) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Aura (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Parosmia (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding the study results for a period up to 30 days from the date the communication is submitted to the sponsor. The sponsor shall have the right to defer proposed publication an additional 60 days from the end of the review period. The sponsor cannot require changes to the communication and cannot unilaterally extend the embargo.